CLINICAL TRIAL: NCT04858321
Title: The Effect of Chronic Passive Heating on Insulin Sensitivity and Cardiovascular Function in People With Type 2 Diabetes Mellitus: A Pre- and Post-test Trial
Brief Title: Chronic Passive Heating in Individuals With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Ant Shepherd, Principal Investigator, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 006
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: We plan to run a within-subject, pre-, post-intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive heating (Experimental): 8-12 x1 h water immersion (to the clavicle, @40 °C, rectal temperature ~38.5 °C and <39 °C) sessions over a period of 14 days.
  Interventions: Procedure: Passive heating

INTERVENTIONS:
Procedure: Passive heating — 8-12 x1 h water immersion (to the clavicle, @40 °C, rectal temperature ~38.5 °C and <39 °C) sessions over a period of 14 days.

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a metabolic condition characterized by chronic hyperglycemia and progressive insulin resistance, which progressively lead to macro- and microvascular damage and subsequent impairments in blood pressure (BP) control. Therapeutic approaches to manage T2DM focus on improving glycaemic control and BP and include pharmaceutical treatments (e.g. Metformin and insulin), physical activity and exercise, and calorie restriction. However, pharmaceutical interventions can be expensive and are associated with low adherence. Although exercise and diet programs have been shown to be effective, like pharmaceutical interventions, they often have poor adherence in people with T2DM. With the number of people with T2DM (464 million) continuing to rise and expected to reach 700 million by 2045, the costs associated with the clinical management of this condition are likely to become unsustainable. There is, therefore, a need to explore the potential of alternative interventions. In particular, interventions which may be cheaper than clinical management and have better adherence than exercise, and hypoglycemic agents, to improve glycemic control and deleterious cardiovascular manifestations of this condition.

Passive heating may be one such intervention with therapeutic potential.

DETAILED DESCRIPTION:
Current estimates suggest 422 million people worldwide live with a form of diabetes, of which ~ 90% have type 2 diabetes mellitus (T2DM). The total direct and indirect cost of care for individuals with diabetes in the UK is £23.7 billion, equating to ~ 20% of the annual NHS budget, this figure is expected to rise to ~£39.8 billion by the year 2035. Approximately 85-90% of cases of T2DM arise from a poor lifestyle and obesity, with the remaining 10-15% resulting from genetic predispositions. Current interventions include pharmaceutical treatments, exercise and calorie restrictive diets, which aim to improve glycaemic control. However, pharmaceutical interventions carry a high financial cost, while exercise and diet programmes have a low adherence rate in individuals with T2DM. With the prevalence of T2DM continuing to increase, the costs associated with the clinical care of these individuals are likely to become unsustainable. Simple, inexpensive interventions to improve the clinical profile of this group are therefore needed.

One emerging potential therapy to improve glucose homoeostasis is passive heating. Preliminary evidence suggests passive heating may have beneficial effects for metabolic health in animal models and in humans. In 1999, the use of hot tubs (38-41°C , 30 mins / day for 3 weeks) was shown to reduce fasting plasma glucose concentrations by ~14% (1.3 mmol.L-1) and decrease HbA1c by ~10-11 mmol/mol in 8 individuals with T2DM. Given the rate of turnover in haemoglobin this reduction is surprising as the treatment period was run over 3 weeks and the total haemoglobin turnover takes ~115 days. While more recent work has been conducted into the effects of a single bout of passive heating in healthy adults and individuals with T2DM (including ourselves, under review), none have been done on chronic heating since Hooper. Hooper postulated that an increase in skeletal muscle blood flow may be responsible for this increased glucose clearance, citing evidence that this can modulate insulin mediated glucose uptake. Other mechanisms have also been purported, but have yet to be elucidated, including; increased insulin sensitivity, altered inflammatory response, activation of heat shock proteins (HSP), altered gut microbiome and butyrate. Repeated passive heating results in transient increases in deep body temperature and may improve glucose homeostasis via similar mechanisms to exercise.

Regular aerobic exercise also improves macro- and microvascular function, muscle oxygenation, autonomic function, cardiorespiratory fitness, lung function and delays age related muscle loss. Acute exercise studies show that insulin sensitivity after 1h of moderate exercise does not change, however, insulin sensitivity appears to be improved following bouts longer than an hour or performed at greater intensity. Increases in insulin sensitivity have a curvilinear relationship with energy expenditure and could also be due to greater HSP expression. However, it is unrealistic for people with T2DM to perform this level of activity. Passive heating may be one supplemental exercise mimetic to augment improvements in insulin sensitivity, cardiorespiratory fitness and muscle strength, and function.

The investigators recently provided evidence that acute passive heating in poeple with T2DM (currently under review for publication) is well tolerated and increases extracellualr [HSP70], and energy expenditure, and reduce diabstolic blood pressure. There is a growing body of evdience that suggests passive heating may improve many facets of human physiology, however, the mechanisms that underpin these benefits have yet to be established and future research needs to explore these further.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (post-menopausal) aged 35 years or above.
* Diagnosed with T2DM as defined by the WHO (≥48 mmol/mol).
* Participant is willing and able to give informed consent for participation in the study.
* Participant is able to understand and fully cooperate with the study protocol.

Exclusion Criteria:

Severe peripheral neuropathy (to the point to which they cannot sense temperature)

* Uncontrolled hypertension (≥180 systolic / 100 diastolic mmHg)
* Taking any medication which may interfere with data interpretation or safety
* Who have had a myocardial infarction or cerebro-vascular event
* Any cardiac abnormalities which restrict hard exercise
* Current smokers or who have stopped within 3 months
* Participant is unable to understand and/or fully cooperate with the study protocol
* Any other serious medical condition which would interfere with data interpretation or safety will be excluded from participation.
* Skin ulcerations
* Eczema
* Pre-existing postural hypertension
* Existing cardiac diseases (identified during screening)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to release IPD, until all avenues of further funding have been exhausted.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-post design, not an RCT. Therefore no assignment details.
Period: Overall Study
Arm/Group | Passive Heating
Started | 17
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14
Height [Mean (Standard Deviation); unit: meters] | 1.68 (0.1)
Mass [Mean (Standard Deviation); unit: kg] | 85 (19)
BMI [Mean (Standard Deviation); unit: kg/m2] | 30 (5.2)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 66 (27)
T2DM duration [Mean (Standard Deviation); unit: years] | 10 (8)
History of microvascular disease [Number; unit: % of cohort] | 21
SBP [Mean (Standard Deviation); unit: mmHg] | 136 (19)
DBP [Mean (Standard Deviation); unit: mmHg] | 81 (11)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Does chronic passive heating improve insulin sensitivity? Calculated using the QUICKI for fasting and Gutt for post-prandial, with glucose and insulin concentrations. A higher value means they have better insulin sensitivity.
Time Frame: Change from pre (day 1) - post 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
AU
  Fasting - pre | 0.31 (0.03)
  Fasting - post | 0.33 (0.04)
  Post-prandial - pre | 0.10 (0.04)
  Post-prandial - post | 0.10 (0.05)

2. Secondary Outcome: Plasma Glucose Concentration
Description: Does chronic passive heating reduce plasma [glucose]?
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
mmol/L
  Fasting - pre | 10.06 (4.51)
  Fasting - post | 9.95 (4.58)
  Post-prandial - pre | 17.34 (7.34)
  Post-prandial - post | 16.84 (6.49)

3. Secondary Outcome: Plasma eHSP70 Concentration
Description: Does chronic passive heating increase plasma [eHSP70]?
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
pg/mL
  Pre | 2435 (984)
  Post | 2524 (790)

4. Secondary Outcome: Plasma IL-6 Concentration
Description: Does chronic passive heating reduce plasma [IL-6]?
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
pg/mL
  Pre | 5.60 (10.46)
  Post | 5.46 (8.47)

5. Secondary Outcome: Plasma IL-10 Concentration
Description: Does chronic passive heating increase plasma [IL-10]?
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
pg/mL
  Pre | 13.55 (35.88)
  Post | 12.50 (31.47)

6. Secondary Outcome: Resting Metabolic Rate
Description: Does chronic passive heating reduce plasma resting metabolic rate?
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
kcal/day
  Pre | 1987 (512)
  Post | 1855 (380)

7. Secondary Outcome: Flow Mediated Dilation
Description: Does chronic passive heating improve macrovascular function? Measured via ultrasound
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: % increase from baseline diameter
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
% increase from baseline diameter
  Pre | 2.88 (1.81)
  Post | 2.45 (1.56)

8. Secondary Outcome: Cutaneous Vascular Conductance
Description: Does chronic passive heating improve microvascular function? Assessed via iontophoresis or the forearm with ACh and Insulin, Area under the curve is the unit. (CVC = skin ﬂux/MAP; ﬂux/mmHg-1)
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: flux/mmHg
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
flux/mmHg
  Insulin AUC - pre | 1.11 (2.10)
  Insulin AUC - post | 0.81 (0.99)
  ACh AUC - pre | 1.52 (1.60)
  ACh AUC - post | 2.06 (2.77)

9. Secondary Outcome: Resting Heart Rate
Description: Does chronic passive heating reduce resting heart rate?
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
beats/min
  Pre | 67 (12)
  Post | 64 (11)

10. Secondary Outcome: Stroke Volume Index
Description: Does chronic passive heating increase stroke volume? Measured noninvasively via thoracic impedance
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
mL/m2
  Pre | 54.6 (13.3)
  Post | 49.4 (11.3)

11. Secondary Outcome: Cardiac Output Index
Description: Does chronic passive heating increase cardiac output? Measured noninvasively via thoracic impedance. L/min/m2 is the unit.
Time Frame: pre - post following 8-12 days of 1 hour of passive heating
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
L/min/m2
  Pre | 3.57 (0.74)
  Post | 3.05 (0.54)

12. Secondary Outcome: TNF-alpha
Description: TNF-alpha
Time Frame: Pre- v post 8-12 1 h hot water immersions
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
pg/mL
  Pre | 10.51 (18.65)
  Post | 10.15 (18.14)

13. Secondary Outcome: Butyric Acid
Description: Butyric acid
Time Frame: Pre- v post 8-12 1 h hot water immersions
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
pg/mL
  Pre | 285 (294)
  Post | 405 (458)

14. Secondary Outcome: SBP
Description: Systolic blood pressure
Time Frame: Pre- v post 8-12 1 h hot water immersions
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
mmHg
  Pre | 136 (19)
  Post | 127 (15)

15. Secondary Outcome: DBP
Description: Diastolic blood pressure
Time Frame: Pre- v post 8-12 1 h hot water immersions
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
mmHg
  Pre | 81 (11)
  Post | 80 (10)

16. Secondary Outcome: MAP
Description: Mean arterial pressure
Time Frame: Pre- v post 8-12 1 h hot water immersions
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
mmHg
  Pre | 99 (11)
  Post | 95 (11)

17. Secondary Outcome: NOX
Description: Nitrates + nitrites
Time Frame: Pre- v post 8-12 1 h hot water immersions
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Passive Heating
Number analyzed (Participants) | 14
micromolar
  Pre | 74.5 (23.7)
  Post | 67.3 (22)

ADVERSE EVENTS:
Time Frame: Approximately 14 days
Arm/Group | Passive Heating
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04858321/Prot_SAP_000.pdf